CLINICAL TRIAL: NCT05405751
Title: Simplified Model of Linkage and Retention to Healthcare System, Using a Mobil Unit and a Same-day Test and Treat Approach Among Excluded Population.
Brief Title: Simplified Model of Linkage and Retention to Care, Using a Mobile Unit and a Same-day Test and Treat Approach Among Excluded Population. (SIMPLIFIED)
Acronym: SIMPLIFIED
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundacion SEIMC-GESIDA (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: GESIDA 12221
Record Dates: First submitted 2022-04-27; First posted 2022-06-06 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2023-07

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — bictegravir; Emtricitabine; tenofovir alafenamide; bictegravir, emtricitabine, tenofovir alafenamide, drug combination

STUDY DESIGN:
Intervention Model Description: Pilot, prospective, single-centre, single-arm, single-treatment study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Patients received BIKTARVY (BIC/FTC/TAF) (Experimental): The patient enrolled in the study and access HIV consulting will start treatment with BIKTARVY the same day of the inclusion. The medication will provided by the sponsor and it will be dispensed by pharmacy service.
  The delivery of medication to the patient can be delegated by a member of investigator staff who pick up the mediaction from pharmacy service to be delivered to the patient. The patient can pick up the medication directly from the pharmacy service. It will be recorded the face to face on delegated dispensing.
  The deliver of medication will be bi-monthly and 2 bottles of tablets will be dispensed. The patients will receive a BIC/FTC/TAF single oral dose per day for 12 months.
  Interventions: Drug: Bictegravir/Emtricitabine/Tenofovir Alafenamide 50 MG-200 MG-25 MG Oral Tablet [BIKTARVY]

INTERVENTIONS:
Drug: Bictegravir/Emtricitabine/Tenofovir Alafenamide 50 MG-200 MG-25 MG Oral Tablet [BIKTARVY] — Patients enrolled in the study and accessing the HIV consultation will start treatment with BIKTARVY on the day of enrollment. Medication will be provided by the sponsor and dispensed through the pharmacy service. The drug will be delivered to the patient with a delegated person outside the hospital environment or it will be the patient himself who picks up the medication.

SUMMARY:
Implementation of a model for access and retention of HIV care for vulnerable and excluded population using a mobile screening unit and a strategy of diagnosis and initiation of treatment with Bictegravir (BIC) 50 mg/ Emtricitabine (FTC) 200 mg / Tenofovir Alafenamide (TAF) 25 mg.

DETAILED DESCRIPTION:
The use of a mobile unit to reach vulnerable HIV-infected people with poor access to the health care system and starting/restarting on the same day ("simplified same day test and treat strategy") is feasible, effective and safe and will allow these people to have a rapid access to ART and long-term follow-up and health care for HIV.

At the screening visit the patient will sign the informed consent form, revise the clinical history and ensure compliance with criteria. A history of drug abuse, complete physical examination, pregnancy test, rapid hepatitis C test, questionnaires and social situation will be collected from the patient.

At the basal visit the patients enrolled in the study will collect lab test (blood count, biochemistry, coagulation, serology, inmunology and virology), vital signs and directed physical examination, concomitant medication and adverse events.

After the basal visit the patient will be followed up on visits week 4, 12, 24, 48 and last visit 50 as follow up safety visit.

ELIGIBILITY:
Inclusion Criteria:

* Vulnerable person ≥18 years
* Understand and sign the informed consent form
* Confirmed HIV infection
* Not receiving ART or on ART with a PVL > copies/ml

Exclusion Criteria:

* Unable to provide contact details
* History of allergy to any of the following drugs: bictegravir, tenofovir alafenamide or emtricitabine
* Taking antiretroviral treatment for less than 1 month
* Pregnancy or breastfeeding at the time of screening or gestational desires during the study period.
* Suspected or diagnosed of active opportinistic disease
* History of severe liver disease (Child- Pugh C) or history of descompensated liver disease (defined as the presence of ascites, encephalopathy, coagulopathy, hypoalbuminaemia, oesophageal or gastric varices or persistent jaundice)
* History of kidney disease CKP-EPI< 30ml/min
* Have any condition that, as per investigator criteria, makes the patient not candidate to be included (active disease, social situation, intoxication...)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-07-04 (Actual); Primary Completion 2023-12-26 (Actual); Study Completion 2024-06-12 (Actual)

PRIMARY OUTCOMES:
To find out whether the implementation of a model of access and retention in care for HIV among vulnerable people using a mobile screening unit and a same-day diagnosis and treatment initiation strategy is effective and safety. | 24-48 weeks
  Proportion of subjects agreeing to participate in the study, proportion of subjects starting ART after inclusion, median time from the study inclusion to ART starting, proportion of subjects with HIV-1 RNA <50 copies/mL at 24 weeks after inclusion, absolute values and changes from baseline in CD4+ cell count and CD4:CD8 at 24 weeks and proportion of subjects making visits at weeks 24 and 48 will be the endponts to measure the effectiveness of the strategy.
  The effectiveness threshold defined is: >80% of enrolled subjects have plasma HIV-1 RNA <50 copies/mL at 24 weeks post-inclusion and who are on follow-up and on ART at remain on follow-up and on ART at week 48.
  Incidence and severity of adverse events (clinical and laboratory) up to 24 weeks, incidence of adverse events leading to discontinuation of treatment up to week 24 and incidence of genotypic resistance mutations in participants with virological failure will be the endpoints to measure the safety of the strategy.

SECONDARY OUTCOMES:
To assess the implementation and feasibility of the intervention | 24-48 weeks
  The evaluation of acceptability, comfort, suitability, usefulness, appropriateness, quality, perceived benefit and satisfaction with the perceived benefit and satisfaction of the intervention at the baseline visit and at the week 24 visit. These parameters will be collected using a scale of 0 to 5 and will be used to measure and assess the implementation of the strategy.
  In addittion to assess the implementation of this project it will be used the endpoints referred to above (Evaluate the effectiveness of the strategy and evaluate the security of the strategy). The time frame for evaluate the effectivebes of the strategy and evaluate the security of the strategy are betwen 24 and 48 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- H. Infanta Leonor, Madrid, Spain